CLINICAL TRIAL: NCT03961490
Title: Contribution of Image Fusion in Percutaneous Left Atrial Occlusion Procedures
Brief Title: Contribution of Image Fusion in Percutaneous Left Atrial Occlusion procédures (Fusion Image)
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0069
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventional study — No interventional study

SUMMARY:
Atrial fibrillation is the most common rhythm disorder, affecting 2 to 3 percent of the population. One of the major complications is the occurrence of thromboembolic events, the thromboembolic risk can be predicted by the ChadsVasc score. Anticoagulant treatment is therefore almost always indicated, however, in view of the target population, anticoagulant treatment is sometimes contraindicated, justifying the appearance of alternative treatment such as occlusion of the left auricle by surgical or percutaneous means, with the placement of a prosthesis in the left auricle.

Image fusion is a new imaging technique aimed at improving the spatial view of 2D images (made during a catheterization session) by repositioning in real time a 3D model obtained by reconstruction from scanner images of the structure of interest. Once the model has been redesigned, it follows all the consequences that the hemodynamicist wants to take and thus guides the gesture as well as possible.

The purpose of this project is to evaluate the contribution of image fusion to per cutaneous occlusion procedures of the left atrium. This contribution will be evaluated by comparing the procedure time, the irradiation time, the amount of contrast material used between the procedures performed with the image fusion technique and without this new technique.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient with a collegially selected indication of FAG
* Patient willing to participate in the study

Exclusion Criteria:

* Minors, adults under guardianship and protected persons
* Presence of contraindications to the procedure, including the presence of a thrombus in the left atrium
* Procedure combined with another percutaneous gesture at the same time

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an elderly population with multiple co-morbidities (hypertension, renal failure, diabetes, etc.), with a major thromboembolic and haemorrhagic risk, and with a formal contraindication to anticoagulant therapy.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
evaluate the contribution of image fusion to reduce patient irradiation with measurement of the amount of irradiation of the procedure | 3 years
  the cumulative Air KERMA in milligray (mGy)
evaluate the contribution of image fusion to reduce patient irradiation with measurement of the amount of irradiation of the procedure | 3 years
  the surface dose product (PDS) in centigray centimetres squared (cGy.cm²)

CONTACTS AND LOCATIONS:
Locations (1):
- Professeur Patrice Guerin, Nantes, France

IPD SHARING:
Plan to Share IPD: No